CLINICAL TRIAL: NCT05614596
Title: Comparative Study Between CT Guided and Fluoroscopic Guided Interventional Techniques for Management of Chronic Low Back Pain
Brief Title: Interventional Techniques for Managment of Chronic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abd El-Rahman Ahmed Omar Salem, Doctor, Assiut University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: chronic low back pain
Record Dates: First submitted 2022-10-14; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CT guided for patient with chronic low back pain (Active Comparator): CT guided treatment in patients with low back pain
  Interventions: Other: CT guided and Flouroscopic guided injection of corticosteroid and local anathesia
- Flouroscopic guided for patient wit chronic low back pain (Active Comparator): Flouroscopic guided treatment in patients with low back pain
  Interventions: Other: CT guided and Flouroscopic guided injection of corticosteroid and local anathesia

INTERVENTIONS:
Other: CT guided and Flouroscopic guided injection of corticosteroid and local anathesia — Patients will be grouped into two groups, the first group (Group A) included patients who were subjected to fluoroscopic guided injection, and the second group (Group B) will include patients who were subjected to CT guided injections.

SUMMARY:
Identify the efficacy of difference procedures of imaging guidance for needles for interventional treatments of low back pain (LBP) associated with sciatica and to study results and satisfaction of the patients between different groups.

DETAILED DESCRIPTION:
Low back pain (LBP) is a major cause of substantial disability. It is usually defined as pain, muscle tension, or stiffness localized below the costal margin and above the inferior gluteal folds, with or without leg pain (sciatica).

Chronic low back pain is defined as the pain that persists for 12 weeks or longer without a response to treatment procedures or the improvement of the underlying cause. Radiculopathy or radicular pain occurs when specific lumbosacral nerve roots are affected, and radicular pain develops due to the irritation of the dorsal root ganglion (DRG). It is characterized by a lumbar pain irradiated to one or more lumbar or sacral dermatomes. Use of fluoroscopy and computed tomography has revolutionized the interventional treatments for chronic low back pain by providing excellent guidance to the needle placement, as well as recognizing improper placements such as intravascular or unintended intrathecal placements of needles and thus avoiding morbidity in the form of injury to the intra-spinal structures including spinal cord, nerve roots and blood vessels. Percutaneous guided interventions such as pulsed radiofrequency (PRF) and transforaminal epidural steroid injection (TFESI) guided by flouroscopy and computed tomography (CT) are safe and effective procedures for the management of chronic RLBP, which can be performed in an outpatient setting without sedation.

Interventional radiologists already possess the technical skills necessary to perform these interventions effectively. Pulsed radiofrequency is one of the interventional therapies for LBP, which uses radiofrequency alternating current to ablate the tissue around the needle electrode. Transforaminal epidural steroid injection (TFESI), as a minimally invasive interventional surgery, is widely used in the treatment of LBP. It has the advantages of less trauma, fewer complications, and faster onset. It relieves symptoms by injecting corticosteroids and local anesthetics around the dural and nerve roots that cause radicular pain.

TFESI combined with PRF for the treatment of RLBP effectively and rapidly relieve radicular pain, reduce VAS (visual analog scale), relieve pain symptoms, improve the quality of life, cure rate, and satisfaction of patients, as well as, achieve long-term remission.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic radicular low back pain with unilateral or bilateral sciatica that persisted for more than 6 months and failed medical treatment for 6 weeks.
2. Pain exacerbates by leaning forward and flexion of the body with numbness and tingling in the legs.
3. Visual analog scale (VAS) of pain severity ≥ 5 related specifically to the daily LBP.
4. Patient develops calf and leg pain of leg raising test.
5. No neurological motor deficits

Exclusion Criteria:

1. Evidance of progressive motor neurological deficits.
2. Magnetic resonance imaging show evidence of > 3 degenerated discs.
3. Intervertebral disc herniation ≥ 4 mm, disc sequestration, extrusion, disc space collapse or spondylolisthesis at the symptomatic level.
4. Moderate to severe central spinal canal or foraminal stenosis
5. Prior lumbar surgery of any kind at the same treatment level
6. Spinal fractures, deformities, infection or tumors.
7. History of uncontrolled coagulopathy or uncontrollable bleeding
8. Patients with psychotic illness, advanced hepatic, uncontrolled diabetic patients.
9. Current pregnancy, recent delivery (within 3-months of consent), or the intent of becoming pregnant during the study period.
10. Local sepsis or skin inflammatory in the back region.
11. Patients with red flags.
12. Neurologic findings (Fecal or urinary incontinence and cauda equina syndrome).
13. Persistent fever (infection).
14. Prolonged use of corticosteroids.
15. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Control of pain by transforaminal epidural steroid injection combined with pulsed radio frequency guided by CT or fluoroscopy | Up to 4 weeks
  Interventional radiologists already possess the technical skills necessary to perform these interventions effectively. Pulsed radiofrequency is one of the interventional therapies for LBP, which uses radiofrequency alternating current to ablate the tissue around the needle electrode. Transforaminal epidural steroid injection (TFESI), as a minimally invasive interventional surgery, is widely used in the treatment of LBP. It has the advantages of less trauma, fewer complications, and faster onset. It relieves symptoms by injecting corticosteroids and local anesthetics around the dural and nerve roots that cause radicular pain.
  TFESI combined with PRF for the treatment of RLBP effectively and rapidly relieve radicular pain, reduce VAS (visual analog scale), relieve pain symptoms, improve the quality of life, cure rate, and satisfaction of patients, as well as, achieve long-term remission.

CONTACTS AND LOCATIONS:
Overall Officials: Faculty Of Medicine, Study Chair — Assiut University
Locations (1):
- Faculty of medicine, Asyut, Egypt